CLINICAL TRIAL: NCT06607926
Title: Efficacy and Safety of Thymosin α1 Plus Immune Checkpoint Inhibitors and Chemotherapy as Neoadjuvant Therapy in Patients With Resectable Stage II - IIIB Non Small Cell Lung Cancer: A Prospective, Multicenter, Randomized, Controlled Trial
Brief Title: Neoadjuvant With Tα1 Plus Immuno-chemotherapy for Resectable NSCLC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, zhang yi, Director of thoracic surgery, Xuanwu Hospital, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XWh-NSCLC-NEO-ZDX
Record Dates: First submitted 2024-09-17; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Resectable Non-Small-Cell Lung Cancer
Keywords: non-small-cell lung cancer; resectable; thymosin alpha-1; PD-1 inhibitor; pCR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Thymalfasin; tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Neoadjuvant therapy with platinum-doublet chemotherapy plus tislelizumab for four cycles, followed by surgery and adjuvant therapy.
  Interventions: Drug: Tislelizumab; Drug: Platinum-doublet chemotherapy
- Experimental group (Experimental): Neoadjuvant therapy with platinum-doublet chemotherapy plus tislelizumab and Tα1 for four cycles, followed by surgery and adjuvant therapy.
  Interventions: Drug: Thymosin Alpha 1; Drug: Tislelizumab; Drug: Platinum-doublet chemotherapy

INTERVENTIONS:
Drug: Thymosin Alpha 1 — 4.8 mg subcutaneous injection twice weekly over 12 weeks
  Other Names: thymalfasin
  Arms: Experimental group
Drug: Tislelizumab — 200mg, IV, d1 of each 21-d cycle, four cycles
Drug: Platinum-doublet chemotherapy — Chemotherapy regimen: (1) for squamous cell carcinoma: cisplatin/carboplatin + paclitaxel; and (2) for non-squamous cell carcinoma: cisplatin/carboplatin + pemetrexed.

SUMMARY:
This study aims to explore the efficacy and safety of thymosin α-1 (Tα1) plus chemotherapy and PD-1 inhibitors as neoadjuvant therapy for operable non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged ≥ 18 years and ≤ 70 years
* With operable NSCLC confirmed by imaging studies and histopathology. (Stage II-IIIB[N2], according to the 8th Edition of the American Joint Committee on Cancer (AJCC-TNM) Staging Manual). Operable NSCLC, as defined by the Multidisciplinary Consensus Statement on the Clinical Management of Patients with Stage III Non-Small Cell Lung Cancer (2019 edition), includes resectable and potentially resectable cases. Resectable stage III NSCLC mainly includes stage IIIA N0-1, N2 with a single mediastinal lymph node metastasis and a short diameter < 2 cm and some T4N1 (with solitary carcinomatous nodules in different lobes of the same lung). Potentially resectable stage III NSCLC includes some IIIA and IIIB tumors, usually including a single N2 mediastinal lymph node with a short diameter < 3 cm, a potentially resectable superior sulcus tumor, and a potentially resectable T3 or T4 central tumor.
* Presence of at least one measurable lesion on imaging as per the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Negative for EGFR and ALK driver mutations
* With an Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 - 1.
* With a life expectancy > 6 months.
* No prior systemic treatment (including surgery, chemotherapy, radiotherapy, targeted therapy, or immunotherapy) for lung cancer.
* Informed consent to undergo radical surgery.
* No contraindications to surgery, as assessed by a thoracic surgeon.
* With adequate organ function, and with laboratory test results meeting the following criteria:

  * Absolute neutrophil count (ANC) ≥ 1.5×10^9/L without the use of granulocyte colony-stimulating factor in the past 14 days
  * Platelet count ≥ 100×10^9/L without blood transfusion in the past 14 days
  * Hemoglobin (Hb) level ≥ 90 g/L without blood transfusion or erythropoietin administration in the past 14 days.
  * Serum creatinine ≤ 1.5 × upper limit of normal (ULN) and creatinine clearance (calculated by the Cockcroft-Gault equation) ≥ 60 mL/min.
  * Total bilirubin ≤ 1.5×ULN; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN.
  * Good coagulation, defined as prothrombin time/international normalized ratio (INR) ≤ 1.5 × ULN.
  * Normal thyroid function, defined as thyroid-stimulating hormone (TSH) level within the reference range. Subjects with baseline TSH level beyond the normal range may also be enrolled if total T3 (or free T3) and free T4 levels are within the normal range.
  * The cardiac enzyme levels are within the normal limits (enrollment is also permitted if the investigator deems laboratory abnormalities as clinically insignificant).
* Females of childbearing potential must agree to use contraceptive methods throughout the study and for 6 months post-study. Patients must have a negative serum or urine pregnancy test within 7 days prior to enrollment and should not be lactating. Male patients must agree to use contraceptive methods throughout the study and for 6 months post-study.
* Subjects have full understanding of the study and voluntarily sign the informed consent form before any trial-related procedure is initiated.

Exclusion Criteria:

* History of other malignancies within 5 years prior to the initial dose, excluding radically treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or carcinoma in situ following radical resection.
* Positive for EGFR and ALK driver mutations or unknown
* Ongoing participation in another interventional clinical trial, or receipt of other investigational agents or devices within 4 weeks prior to the first dose.
* Prior multidisciplinary treatment for lung cancer, including but not limited to surgery, radiotherapy, chemotherapy, and/or immunotherapy (e.g., PD-1 or PD-L1 inhibitors and CTLA-4 inhibitors).
* Use of systemic therapy with anti-tumor traditional Chinese patent medicines or immunomodulatory drugs (including thymopeptides, interferons, and interleukins, except for topical use for pleural effusions) within 2 weeks before the first dose.
* Active autoimmune disease necessitating systemic treatment (e.g., disease-modifying drugs, glucocorticoids, and immunosuppressants) within 2 years before the first dose. Replacement therapies such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency are not classified as systemic therapy.
* Use of systemic glucocorticoid therapy (excluding intranasal, inhaled, or other topical applications) or any other immunosuppressive treatment within 7 days before the first dose. Note: Glucocorticoids at physiological doses (≤ 10 mg/day of prednisone or equivalent) are allowed.
* History of allogeneic organ transplantation (excluding corneal transplantation) or allogeneic hematopoietic stem cell transplantation.
* Allergic to the active substance or excipients of the study drug.
* Incomplete recovery from toxicity and/or complications due to prior interventions (i.e., ≤ grade 1 or baseline, excluding fatigue and alopecia) before treatment initiation.
* Known history of human immunodeficiency virus (HIV) infection (i.e., positive for HIV-1/2 antibody).
* Untreated active hepatitis B, defined as positive HBsAg along with HBV-DNA levels exceeding the ULN as determined by the clinical laboratory of the research center. Note: Subjects with hepatitis B may be eligible if they meet the following criteria:

  * The HBV viral load is < 1000 copies/mL (200 IU/mL) before the first dose, with subjects being required to undergo anti-HBV therapy throughout chemotherapy to prevent viral reactivation.
  * For subjects with anti-HBc(+), HBsAg(-), anti-HBs(-), and HBV viral load (-), no HBV prophylaxis is required, although viral reactivation should be monitored closely.
* Subjects with active hepatitis C virus (HCV) infection, defined as positive HCV antibody and HCV-RNA levels above the threshold of detection.
* Administration of a live vaccine within 30 days before the first dose. Note: administration of inactivated influenza vaccine by injection within 30 days before the first dose is allowed; however, subjects with a history of administration of intranasal live attenuated influenza vaccines will be excluded.
* Pregnant or lactating women.
* Subjects with any severe or uncontrolled systemic condition, including but not limited to:

  * Significant resting ECG abnormalities in rhythm, conduction, or morphology (e.g., complete left bundle branch block, second- and higher-degree heart block, ventricular arrhythmias, or atrial fibrillation), corresponding to severe and difficult-to-control symptoms.
  * Unstable angina, congestive heart failure, or New York Heart Association (NYHA) class ≥ 2 chronic heart failure.
  * History of arterial thrombosis, embolism, or ischemia, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, within 6 months preceding enrollment.
  * Uncontrolled blood pressure, with systolic blood pressure (SBP) > 140 mmHg or diastolic blood pressure (DBP) > 90 mmHg.
  * History of non-infectious pneumonitis necessitating glucocorticoid therapy within 1 year before the first dose, or current clinically active interstitial lung disease.
  * Active tuberculosis.
  * Active or uncontrolled infection requiring systemic treatment.
  * Clinically active diverticulitis, intra-abdominal abscess, or gastrointestinal obstruction.
  * Liver diseases, including cirrhosis, decompensated liver disease, and acute/chronic active hepatitis.
  * Poorly controlled diabetes mellitus, with fasting blood glucose (FBG) > 10 mmol/L.
  * Urine protein ≥++ on routine urinalysis, along with a 24-hour urine protein level of > 1.0 g.
  * A psychiatric disorder that limits the patient's ability to comply with the treatment or to follow the protocol.
* A history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study; or, any condition that is judged by the Investigator to be inappropriate for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate | at the time of surgey
  The rate of no viable tumor cells in the resected specimen including lymph node region evaluated by H&E staining

SECONDARY OUTCOMES:
major pathological response rate | at the time of surgey
  The rate of ≤ 10% viable tumor cells in the resected specimen evaluated by H&E staining
Rate of R0 resection | at the time of surgey
  The rate of participants undergoing R0 resection
Incidence of irAE | From the first dose of PD-1 inhibitors to the three months after surgery
  The occurrence rate of immune-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, Study Director — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No